CLINICAL TRIAL: NCT06179953
Title: Evaluate the Effect of Social Robot Mediation on the Development of Emotional Skills
Brief Title: Emotional Skills Training with Social Robot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2023-010
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; children; emotional skills; social robot
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group with social robot (Experimental): The emotional skills protocol aims to achieve the following objectives:
  * Acquisition of appropriate emotional skills and understanding of emotions;
  * Construction of functional thoughts related to emotions;
  * Enhancement of interpersonal and social skills. It is aimed at a sample of children diagnosed with high-functioning autism spectrum disorder (ASD) between the ages of 5 and 10. The experimental group will carry out training through the use of social robots. The robot provides instructions and if the child requests it, it gives prompts.
  Interventions: Other: NAO intervention
- Control group without social robot (Other): The emotional skills protocol aims to achieve the following objectives:
  * Acquisition of appropriate emotional skills and understanding of emotions; Construction of functional thoughts related to emotions;
  * Enhancement of interpersonal and social skills. It is aimed at a sample of children diagnosed with high-functioning autism spectrum disorder (ASD) between the ages of 5 and 10. Control group which will be conducted through traditional therapy. The therapist provides instructions, and if the child has difficulty responding, he gives prompts.
  Interventions: Other: Traditional intervention

INTERVENTIONS:
Other: NAO intervention — The protocol is divided into 4 stages:
  1. EMOTION RECOGNITION - "Mime Game": activity aimed at acquiring the ability to label basic emotions.
  2. EMOTION/SITUATION ASSOCIATION - "How do I feel when...?" game: presentation of social situations to acquire the ability to attribute the emotion associated with the situation presented.
  3. DIFFERENTIATION BETWEEN EMOTIONS AND THOUGHTS - "Think-Feel Game": activity aimed at differentiating thoughts from emotions and acquiring the skill of linking a thought to an emotion.
  4. LEARNING A REPERTOIRE OF USEFUL THOUGHTS: acquisition of useful thoughts related to certain emotional situations. The robot provides instructions and if the child requests it, it elects prompts.
  Arms: Experimental group with social robot
Other: Traditional intervention — The protocol is divided into 4 stages:
  1. EMOTION RECOGNITION - "Mime Game": activity aimed at acquiring the ability to label basic emotions.
  2. EMOTION/SITUATION ASSOCIATION - "How do I feel when...?" game: presentation of social situations to acquire the ability to attribute the emotion associated with the situation presented.
  3. DIFFERENTIATION BETWEEN EMOTIONS AND THOUGHTS - "Think-Feel Game": activity aimed at differentiating thoughts from emotions and acquiring the skill of linking a thought to an emotion.
  4. LEARNING A REPERTOIRE OF USEFUL THOUGHTS: acquisition of useful thoughts related to certain emotional situations. The therapist provides instructions, and if the child has difficulty responding, he or she may ask the operator for prompts.
  Arms: Control group without social robot

SUMMARY:
Autism is a neurodevelopmental disorder that involves difficulties especially in the sphere of social interaction, social communication, and restricted and stereotyped behavior patterns.

In particular, emotional regulation is a central developmental skill. In fact, the emotional dysregulation observed in children with autism results in increased social and behavioral difficulties over time.

Therefore, the present protocol aims to test the role of a human-assisted social robot as a mediator of social-emotional understanding intervention for children with autism spectrum disorders (ASD).

The children, will be divided into two groups, an experimental one in which training will be conducted through the use of social robot and control group which will be conducted through traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Language in sentences
* use of connectors
* ability to narrate events not present
* ADOS level: module 2
* Griffiths: QS>75

Exclusion Criteria:

* presence of other medical disorders

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Test of Emotional Vocabulary | The administration has a duration of 15 minutes.
  The Test of Emotional Vocabulary contains an initial board, with which the child is introduced to the two protagonists of the subsequent stories, a boy and a girl; there is then a pretest board and 14 storyboards. For each of them, the examiner reads the short story to the child and then asks the child to choose, from two alternative emotional words, the one that best expresses what the protagonist of the story is feeling. In the first part, the child's understanding of emotional vocabulary referring to six basic emotions plus one complex emotion (joy, happiness, sadness, anger, fear, disgust and shame) is assessed; in the second part, the emotional terms all refer to complex emotions (guilt, envy, jealousy, contempt, hate, longing and pride).
Test of emotion comprehension | The administration has a duration of 15-20 minutes.
  The Test of emotion comprehension (TEC) is an instrument to assess a child's understanding of emotions, in its various aspects, that is, the nature, causes, and ways of controlling and regulating emotions. It is used for children aged 3-4 to 10-11 years. It is administered by telling a story in pictures, the child responds by indicating and finally, it takes about 15-20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.) https://doi.org/10.1176/appi.books.9780890425596.
- [Background] Berkovits, L., Eisenhower, A. e Blacher, J. (2017). Regolazione delle emozioni nei bambini piccoli con disturbi dello spettro autistico. Giornale di autismo e disturbi dello sviluppo, 47(1), 68-79.